CLINICAL TRIAL: NCT00234910
Title: A Phase III, Open Label, Randomized, Comparative Study of the Antiviral Efficacy of ARV Therapy With Lopinavir/Ritonavir (LPV/r-Kaletra) in Combination With Tenofovir (TDF) Versus Standard of Care (Kaletra in Combination With 2 Nucleoside RTIs) in naïve-HIV-1 Positive Patients
Brief Title: Efficacy of Simplified Two Drug Kaletra Regimen vs. Kaletra Triple Drug Standard of Care Regimen in Treatment naïve HIV Infected Patients
Acronym: KALEAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Dr. Umberto di Luzio Paparatti, Medical Director Abbott Italy, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITAL-04-002; EUDRACT 2004-000786-35; KALEAD
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: HIV Infection
Keywords: Lopinavir; Ritonavir; Kaletra; Tenofovir; HIV infection; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 2 drug arm
  Interventions: Drug: Tenofovir DF; Drug: lopinavir/ritonavir with 2 Nucleoside RTIs
- B (Active Comparator): 3 drug arm, SOC
  Interventions: Drug: lopinavir/ritonavir with 2 Nucleoside RTIs

INTERVENTIONS:
Drug: Tenofovir DF — TDF 300mg QD for 72 wks
  Arms: A
Drug: lopinavir/ritonavir with 2 Nucleoside RTIs — LPV/rSGC 400/100mg BID + 2 nucleoside RTIs as prescribed by the Investigator for 72 wks
  Other Names: ABT-378; Kaletra; lopinavir/ritonavir

SUMMARY:
The purpose of this study is to obtain a preliminary assessment of the antiviral activity and tolerability of simplified Kaletra dual agent therapy as initial treatment for HIV infection, relative to a Kaletra three drug standard of care reference arm.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* >18 years of age
* HIV RNA> 400 copies/mL
* Any CD 4 cell count
* Antiretroviral naïve
* No acute illness

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Antiviral efficacy by HIV RNA | 72 wks
Incidence of adverse events | 72 wks

SECONDARY OUTCOMES:
Adherence and quality of life | 72 wks

CONTACTS AND LOCATIONS:
Overall Officials: Umberto di Luzio Paparatti, MD, Study Director — Abbott
Locations (1):
- Global Medical Information-Abbott, Abbott Park, Illinois, United States